CLINICAL TRIAL: NCT05352048
Title: Prospective Evaluation of Mechanomyography Versus Triggered Electromyography for Intraoperative Assessment of Cortical Breaches During Instrumented Lumbar Spine Surgery
Brief Title: MMG vs. EMG for Cortical Breach Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francis Farhadi (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor-Investigator, Francis Farhadi, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 76122
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Low Back Disorder
Keywords: Lower back surgery; Lumbar fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intraoperative MMG vs EMG for cortical breach detection (Experimental): Participants in this arm will be assessed with both MMG and EMG during their lower spine fusion surgery.
  Interventions: Device: Triggered Electromyography; Device: Mechanomyography

INTERVENTIONS:
Device: Triggered Electromyography — Triggered electromyography will be used during surgery to detect nerve impingement by pedicle screws used for spinal fusion. Threshold stimulation data from the device will be recorded.
Device: Mechanomyography — SENTIO MMG ball tip probe will be used during surgery to detect nerve impingement by pedicle screws used for spinal fusion. Threshold stimulation data from the device will be recorded, and the accuracy compared to the data from the triggered electromyography.
  Other Names: SENTIO MMG

SUMMARY:
The purpose of this study is to determine how well mechanomyography (MMG) and electromyography (EMG) prevent cortical bone breaches, or the pinching of a nerve from screw placement, in patients having lower back surgery requiring hardware. Both MMG and EMG are devices approved by the FDA to detect the location of nerves during surgery so they can be avoided. The results from both tests will be compared to one another to determine if one is better at accurately locating nerves than the other.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo a one-, two-, or three-level posterolateral spinal fusion surgery using Depuy Synthes Expedium pedicle screw instrumentation.
* over the age of 18 years old
* unresponsive to conservative care for a minimum of 6 months
* psychosocially, mentally, and physically able to fully consent and comply with this protocol

Exclusion Criteria:

* preexisting medical condition or comorbidity that makes them a poor candidate
* open wound local to the operative area, or rapid joint disease, bone absorption, or osteoporosis
* requires medications that may interfere with bone or soft tissue healing
* active local or systemic infection
* metal sensitivity/foreign body sensitivity
* implanted pacemaker
* morbidly obese, defined as a body mass index (BMI) greater than 45
* osteoporosis
* involved in or planning to engage in litigation or receiving Workers Compensation related to neck or back pain.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Francis Farhadi, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraoperative MMG vs EMG for Cortical Breach Detection
Started | 65
Completed | 61
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — did not get EMG-MMG readings intraoperatively | 3

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative MMG vs EMG for Cortical Breach Detection
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.26 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 59
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Success of Pedicle Screw Trajectories
Description: Patients with successful pedicle screw trajectories determined by the percentage of patients with A/B or C/D/E breaches.
  * Grade A - No cortical breach (0 mm)
  * Grade B - Pedicle cortical breach < 2 mm
  * Grade C - Pedicle cortical breach = 2 to < 4 mm
  * Grade D - Pedicle cortical breach = 4 to < 6 mm
  * Grade E - Pedicle cortical breach = 6 mm
Time Frame: 1 hour
Measure: Count of Units; unit: Screws
Units Other Than Participants: Screws
Arm/Group | Intraoperative MMG vs EMG for Cortical Breach Detection
Number analyzed (Participants) | 61
Number analyzed (Screws) | 303
Screws
  Grade A or B | 296
  Grade C | 5
  Grade E | 2

2. Secondary Outcome: Change From Baseline in the Numeric Rating Scale (NRS) Questionnaire for Pain.
Description: This survey is used to assess pain experienced by the subject and the severity of the pain. Types of pain include numbness, pins and needles, dull aching, burning sensation, muscle cramps, and stabbing pain. Pain severity is rated on a scale of 0-10 where 0 is no pain and 10 is the worst pain imaginable. Pain is assessed in the back and legs. Changes reported as percentages using the formula [(Average measure at 3 months - Average measure at baseline)/Average measure at baseline].
Time Frame: 3 months after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intraoperative MMG vs EMG for Cortical Breach Detection
Number analyzed (Participants) | 61
score on a scale
  NRS Back Pain | -3.80 (3.22)
  NRS Leg Pain | -4.15 (3.41)

3. Secondary Outcome: Change From Baseline in the Oswestry Disability Index Version 2.1A
Description: This survey is used to quantify disability for low back pain. There are five disability categories ranging from minimally disabled to crippled. The appropriate disability category is determined by the sum of the subjects points divided by the total possible points(50) times 100. This yields a % disabled score and this % determines the appropriate category designation. 0% is equated with no disability and 100% is the maximum disability possible. Changes reported as percentages using the formula [(Average measure at 3 months - Average measure at baseline)/Average measure at baseline]
Time Frame: 3 months after surgery
Measure: Mean (Standard Deviation); unit: percentage of disability
Arm/Group | Intraoperative MMG vs EMG for Cortical Breach Detection
Number analyzed (Participants) | 61
percentage of disability | -47.4 (34.2)

4. Secondary Outcome: Change From Baseline in the PROMIS Global-10
Description: This questionnaire is a 10 item patient reported tool used to quantify the patients general healthcare related quality of life. It assesses both physical and mental health and is scored as a percentage. Scores closer to 100% report a better quality of life than those who score lower. Changes reported as percentages using the formula [(Average measure at 3 months - Average measure at baseline)/Average measure at baseline]
Time Frame: 3 months after surgery
Measure: Mean (Standard Deviation); unit: percentage of quality of life
Arm/Group | Intraoperative MMG vs EMG for Cortical Breach Detection
Number analyzed (Participants) | 61
percentage of quality of life
  Physical Health | 26.6 (38)
  Mental Health | 14.6 (28)

5. Secondary Outcome: Change in the Short-From (SF-36) Health Survey
Description: This survey quantifies how a patient feels about their health, and how well they are able to do common activities. This survey has 9 domains that assess the patients functional ability. The domains are scored as percentages from 0%-100% with 0% being severely limited and 100% being no deficits.
Time Frame: 6 weeks and 3 months after surgery
Population: Survey data never collected due to redundancy and overlapping questions contained in the PROMIS-10 survey.
Arm/Group | Intraoperative MMG vs EMG for Cortical Breach Detection
Number analyzed (Participants) | 0

6. Secondary Outcome: Hospital Readmission at 30 Days
Description: Percent of patients undergoing hospital readmission 30 days following the procedure.
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative MMG vs EMG for Cortical Breach Detection
Number analyzed (Participants) | 61
percentage of participants | 3.28

7. Secondary Outcome: Hospital Readmission at 90 Days
Description: Percent of patients undergoing hospital readmission 90 days following the procedure.
Time Frame: 90 days
Measure: Number; unit: Percentage of participants
Arm/Group | Intraoperative MMG vs EMG for Cortical Breach Detection
Number analyzed (Participants) | 61
Percentage of participants | 1.64

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Intraoperative MMG vs EMG for Cortical Breach Detection
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 3/61
Other Adverse Events (participants affected / at risk) | 23/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative MMG vs EMG for Cortical Breach Detection (N=61)
ankle fracture (Musculoskeletal and connective tissue disorders) | 1
Lower extremity deep venous thrombosis (Blood and lymphatic system disorders) | 1
Stroke (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative MMG vs EMG for Cortical Breach Detection (N=61)
Upper Limb Swelling (Blood and lymphatic system disorders) | 1
Low hemoglobin (Blood and lymphatic system disorders) | 1
Postoperative anemia (Blood and lymphatic system disorders) | 1
Hypotension (Cardiac disorders) | 1
Left eye pain (Eye disorders) | 1
Bowel Impaction (Gastrointestinal disorders) | 1
Postoperative ileus (Gastrointestinal disorders) | 1
Mechanical Fall (General disorders) | 3
Tooth Abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Suture abscess (Infections and infestations) | 1
High fasting blood glucose (Metabolism and nutrition disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Right foot drop (Nervous system disorders) | 1
Postoperative foot drop (Nervous system disorders) | 1
Left sided sciatic pain (Nervous system disorders) | 1
Superficial wound dehiscence (Surgical and medical procedures) | 2
Wound dehiscence (Surgical and medical procedures) | 1
Intraoperative CSF leak (Surgical and medical procedures) | 1
Posterior tibial vein deep venous thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-12-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT05352048/Prot_SAP_ICF_001.pdf